CLINICAL TRIAL: NCT03314051
Title: Long-term Treatment Outcome for Stage III Nasopharyngeal Carcinoma Patients and Risk Grouping by Plasma Epstein-Barr Virus DNA
Brief Title: Long-term Treatment Outcome for Stage III NPC Patients and Risk Grouping by Plasma EBV DNA
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE12117
Record Dates: First submitted 2017-10-15; First posted 2017-10-19 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Nasopharyngeal Carcinoma; EBV Related Carcinoma
Keywords: Nasopharyngeal Carcinoma; plasma EBV DNA
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — We collected the pre-treatment and post-treatment plasma EBV DNA. The plasma EBV DNA assay was analyzed by real time PCR.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
No previous study reported the treatment outcome of stage III nasopharyngeal carcinoma (NPC) patients. The investigators try to investigate the long-term treatment outcome of stage III NPC patients and do risk grouping by plasma Epstein-Barr virus (EBV) DNA assay for future therapy improvement.

DETAILED DESCRIPTION:
The stage III NPC patients were the majority group of the patient population of NPC. But most clinical trials focused on the treatment of American Joint Committee on Cancer (AJCC) 7th edition stage IVA/IVB treatment for high risk of recurrence or metastasis. No previous study reported the treatment outcome of stage III NPC patients. The investigators tried to investigate the long-term treatment outcome of stage III NPC patients and do risk grouping by plasma EBV DNA assay for future therapy improvement.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven stage III nasopharyngeal carcinoma (NPC)
* Finished curative chemoradiotherapy
* Have Pre-treatment and post-radiotherapy plasma EBV DNA

Exclusion Criteria:

* No tissue proven NPC
* Not finished curative treatment
* No Pre-treatment and post- radiotherapy plasma EBV DNA

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tissue proven stage III NPC patients and received curative treatment in our institute. Pre-treatment and post-radiotherapy plasma EBV DNA will be obtained.
Sampling Method: Probability Sample
Enrollment: 366 (Actual)
Dates: Start 2012-05-02 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 5 year
  Diagnosis to death

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 5 year
  Diagnosis to death to recurrence or metastasis
Distant metastasis failure-free survival (DMFFS) | 5 year
  Diagnosis to death to distant metastasis
Locoregional failure-free survival (LRFFS) | 5 year
  Diagnosis to death to locoregional failure

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ching Lin, MD.PhD., Principal Investigator — Department of Radiation Oncology, Taichung Veterans General Hospital